CLINICAL TRIAL: NCT00142961
Title: Marijuana-Abusing Attention Deficit Hyperactivity Disorder (ADHD) Teens: Atomoxetine Treatment
Brief Title: Atomoxetine for Treating Marijuana-Abusing Adolescents Who Have Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #4988-NIDA-19233-1; R01DA019233 (NIH); DPMCDA
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Marijuana Abuse
Keywords: cannabis abuse; atomoxetine; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Marijuana Abuse | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Atomoxetine prescribed daily
  Interventions: Drug: Atomoxetine
- 2 (Placebo Comparator): placebo controlled arm
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Atomoxetine — atomoxetine
  Arms: 1
Other: placebo
  Arms: 2

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is common among adolescents seeking treatment for marijuana dependence. The purpose of this study is to determine the use of atomoxetine in treating adolescents who abuse marijuana and have ADHD. In addition, this study will assess whether atomoxetine reduces ADHD symptoms as compared to a placebo. Finally, the study will determine whether atomoxetine improves treatment retention and progress in adolescents with ADHD and marijuana dependence.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is common among adolescents seeking treatment for marijuana dependence. Therefore, it is important to develop treatments targeting adolescents diagnosed with both ADHD and marijuana dependence. Atomoxetine is currently used to treat individuals diagnosed with ADHD. The purpose of this study is to determine the feasibility of administering atomoxetine in a therapeutic setting to adolescents who abuse marijuana and have ADHD. In addition, this study will assess whether atomoxetine reduces ADHD symptoms. Finally, this study will determine whether atomoxetine improves treatment retention and progress in adolescents with ADHD and marijuana dependence.

Participants in this double-blind study will be randomly assigned to receive either atomoxetine or placebo. Study visits will occur 2 times each week for the duration of the 12-week trial. At each study visit, vital signs and medication side effects will be assessed. In addition, psychiatric ratings measurements will be evaluated. Participants will also complete self reports in order to track ADHD-related symptoms. Starting at the Week 2 study visit, all participants will receive psychotherapy sessions. This will involve cognitive-behavioral therapy/relapse prevention treatment that has been designed specifically for ADHD adolescents. The aim of the cognitive skills training will be to assist the participants in developing the skills necessary to manage their drug use as well as the symptoms they experience related to ADHD. At Month 6, a follow-up visit will occur, at which time participants urine toxicology tests will be completed to determine if participants have been using marijuana or any other substances of abuse. In addition, at the Month 6 follow-up visit, participants will complete psychiatric ratings, self reports, and will meet with a physician to assess ADHD-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for marijuana dependence and reports that marijuana is their primary drug of abuse
* Meets DSM-IV criteria for ADHD, as determined by the CAADID
* Females will be included if not pregnant or breastfeeding, and agree to use an adequate method of contraception for the duration of the study

Exclusion Criteria:

* Meets DSM-IV criteria for schizophrenia, schizoaffective illness, psychotic disorder other than transient psychosis due to drug abuse, current major depression, bipolar illness, or psychiatric disorders (individuals with substance-induced mood disorder with depressive features as well as substance induced anxiety disorder will not be excluded from the study)
* Medically unstable (based on laboratory tests, an electrocardiogram, medical history, and physical examination) such that study participation would be hazardous; examples include uncontrolled high blood pressure and faster than normal heart rate (systolic blood pressure greater than 130, diastolic blood pressure greater than 80, or a resting heart rate greater than 90) or diabetes
* History of seizures
* Current suicidal risk
* Pregnant or breastfeeding
* Physiologically dependent on any other drugs (excluding nicotine) that requires a medical intervention
* Known sensitivity to atomoxetine
* Prior treatment failure with atomoxetine
* Currently receiving effective treatment with atomoxetine
* Coronary vascular disease, as indicated by a history or suspected by an abnormal ECG or history of cardiac symptoms
* Currently taking a psychotropic medication
* Currently taking cough medicine (e.g., dextromethorphan) or albuterol
* Currently taking or history of taking monoamine oxidase inhibitors (MAOIs) within 2 weeks prior to enrollment
* Narrow angle glaucoma
* Hepatitis
* Adolescents who are prisoners as defined by OHRP regulations, namely directly court-mandated adolescents (as opposed to probation or parole-mandated clients, as well as voluntary clients, who will not be excluded)

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
ADHD response and reduction in ADHD symptoms; measured at Week 12 | 12 weeks of trial or length of participation

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Phoenix House, New York, New York, United States

REFERENCES:
- See also: Substance Treatment and Research Service — http://www.stars.columbia.edu